CLINICAL TRIAL: NCT04495023
Title: Left Elective Colectomy in Renal Transplanted Patients : a Case-control Study (LECoRT Study)
Brief Title: Left Elective Colectomy in Renal Transplanted Patients
Acronym: LECoRT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Department of Visceral and Digestive Surgery, Centre hospitalier de Dunkerque (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0356
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-07

CONDITIONS: Left Elective Colectomy; Renal Transplanted Patients
Keywords: Benign or malign pathology; Renal transplanted patients; Anastomotic leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Kidney transplanted patients): Group 1: Kidney transplanted patients requiring oncologic or non-oncologic left elective colectomy All kidney transplanted patients requiring oncologic or non-oncologic left elective colectomy between 01 January 2004 and 31 December 2015.
  Interventions: Procedure: Left elective colectomy
- Group 2 (Non-transplanted patients): Group 2 : Non-transplanted patients requiring oncologic or non-oncologic left elective colectomy Non-transplanted patients requiring oncologic or non-oncologic left elective colectomy between 01 January 2004 and 31 December 2015.
  Interventions: Procedure: Left elective colectomy

INTERVENTIONS:
Procedure: Left elective colectomy — Open or laparoscopic left elective colectomy with colo-rectal anastomosis

SUMMARY:
Aim of the study :

To evaluate postoperative outcomes of elective left-sided colectomy in a renal transplanted population.

Methods :

From 2010 to 2015, all consecutive patients who underwent left elective colectomy in a referral center were prospectively collected.

Considering our exclusion criterial, data from 120 patients were analyzed. The cohort was separated into 2 groups : renal transplanted patients (KTR-group) and non-renal transplanted patients (C-group) Short and longterm outcomes were compared between the two groups.

Primary outcome :

90 days postoperative anastomotic leak rate

DETAILED DESCRIPTION:
From January 2010 to December 2015, data from patients requiring an elective left colectomy for benign or malignant indication were collected prospectively in our colorectal surgery database.

According to our exclusion criterial patients were retrospectively divided into two groups: kidney transplant recipients (KTR-group) and control group (C-group).

The surgical indication for an oncologic left colectomy was retained by the expert surgeon, after a multidisciplinary conversation meeting comprising at least one surgeon, one gastroenterologist, one nephrologist, one radiologist and one oncologist. The surgical indication for diverticular disease was based on French guidelines.

Demographic, clinical, intraoperative and postoperative, histological, length of hospital stay and mortality data were collected over a 90-day period following the intervention.

ELIGIBILITY:
Inclusion criteria:

* Open or laparoscopic left elective colectomy with colo-rectal anastomosis
* age > 18 y.o.

Exclusion criteria:

* emergency surgery
* past history of rectal surgery
* ASA I

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who Open or laparoscopic left elective colectomy with colo-rectal anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of Anastomotic leak after left elective colectomy | 90 days postoperative
  Anastomotic leak according to the International Study Group of Rectal Cancer

SECONDARY OUTCOMES:
Long term outcomes | 1 day
  Status at the date of latest news

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Bardol T, Souche R, Genet D, Ferrandis C, Guillon F, Pirlet I, Fabre JM. Outcomes of elective left colectomy in renal-transplanted patients: a single-center case-control study (LECoRT study). Int J Colorectal Dis. 2021 Jun;36(6):1209-1219. doi: 10.1007/s00384-021-03860-7. Epub 2021 Jan 28. PMID 33511479